CLINICAL TRIAL: NCT06583590
Title: Evaluation of Efficacy of Botulinum Toxin A Plus Oral Tadalafil 5 mg in Diabetic Men With Erectile Dysfunction Not Responding to Approved Oral or Intracorporeal Vasoactive Treatments.
Brief Title: Evaluation of Efficacy of Botulinum Toxin A Plus Oral Tadalafil 5 mg in Diabetic Men With Erectile Dysfunction
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Aswan University Hospital (Other)
Collaborators: Aswan University (Other); Cairo University (Other)
Responsible Party: Principal Investigator, El Hassan Mohsen Mansour Mahmoud, Assistant lecturer, Aswan University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 943/7/24
Record Dates: First submitted 2024-08-09; First posted 2024-09-04 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Erectile Dysfunction With Diabetes Mellitus
MeSH Terms: interventions — Botulinum Toxins, Type A; Tadalafil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group 1 (Other): 32 patients will be injected single intracavernosal injection of 100 unit of Botulinum toxin A accompained by oral daily tadalafil 5 mg for 3 months.
  Interventions: Drug: Botulinum toxin A; Drug: Tadalafil 5mg

INTERVENTIONS:
Drug: Botulinum toxin A — Botulinum toxin (BoNT) is One of the most potent toxins known to humans produced by Clostridium botulinum that has been used to treat several striated and smooth muscle disorders. Because the pathophysiology and the reason for patients' lack of response to PDE5I is insufficient smooth muscle relaxation and veno-occlusive disorder (VOD) , BTX-A may prove to be a viable treatment for this patient population due to its availability to facilitate long-acting cavernosal smooth muscle relaxation by inhibition of the release of noradrenaline from the adrenergic neurons acting on the cavernosal smooth muscle. Thus, the dominant sympathetic basal tone of the cavernosal smooth muscle is essentially removed, facilitating the occurrence of an erection.
  Other Names: Botox; BTX-A
Drug: Tadalafil 5mg — Tadalafil is one of 5-phosphodiesterase inhibitors that used to treat male sexual function problems (impotence or erectile dysfunction-ED). In combination with sexual stimulation, tadalafil works by increasing blood flow to the penis to help a man get and keep an erection.Tadalafil is also used to treat the symptoms of an enlarged prostate (benign prostatic hyperplasia-BPH). It helps to relieve symptoms of BPH such as difficulty in beginning the flow of urine, weak stream, and the need to urinate often or urgently (including during the middle of the night). Tadalafil is thought to work by relaxing the smooth muscle in the prostate and bladder.

SUMMARY:
Study is aiming to evaluate safety, efficacy and durability of intracavernosal injection (ICI) of Botulinum toxin A plus oral tadalafil in controlled diabetic men with refractory Erectile Dysfunction.

DETAILED DESCRIPTION:
Total of (32) male patients will be included in this study and will be recruited from the Andrology, Sexology & STDs outpatient clinics- Faculty of medicine -Cairo and Aswan Universities. All those patients are complaining of erectile dysfunction Unresponsive to Approved Pharmacological Treatments. Each patient will have an informed consent obtained prior to conducting the study.

All patients will be subjected to the following:

* History taking.
* Clinical examination (general and local genital examination).
* International Index of Erectile Function (IIEF-5) before and after treatment (Rosen et al., 2002).
* Erection Hardness Score (EHS) before and after treatment (Mulhall et al., 2006).
* Global assessment questionnaire after treatment (Giuliano et al., 2007).

  * All patients will be examined by Duplex Doppler ultrasonography in the basal condition and after the induction of penile erection with the assistance of an intracavernous injection of alprostadil 20 μg/mL.
  * All patients will receive single dose of ICI of 100u of (BTXA) combined with 5mg oral Tadalafil once daily for 3 months.
  * The subjects will be re-examined and International Index of Erectile Function (IIEF-5), Erection Hardness Score (EHS)and penile color Doppler ultrasound with PGE-1 injection will be done at 6 and 12 weeks from the start of therapy in addition to Global assessment questionnaire will be done at 12 weeks from the start of therapy

    * Procedure
  * The patients will lied down in supine position. After cleansing the skin with alcohol, intracavernosal injection of single dose 100U (BTX-A) diluted in isotonic saline 2cm proximal to coronal margin at right and left sides will be performed and the injection site will be pressed directly for two minutes. To prevent systemic toxicity, a veno-occlusive ring will be used at the base of the penis at the time of injection and will be kept in place for 15 minutes after injection.

ELIGIBILITY:
Inclusion Criteria:

* Adult controlled diabetic married men who proved to be vasculogenic ED by Penile Duplex.
* Men who had shown an insufficient response for at least 3 months to the registered PDE5-Is at the highest approved dose, either on-demand or daily, or to PGE1 ICIs.
* Severe erectile dysfunction (erection hardness score ≤ E3 after intracavernosal injection of PGE-1).

Exclusion Criteria:

* Men who had cardiovascular disease interfering with sexual activity.
* Men with history of an unstable psychiatric conditions
* Presence of penile anatomical abnormalities that would significantly impair erectile function.
* History of spinal or pelvic radical surgery.

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Treatment. | 3 months
  The primary outcome is to assess the effect of single intra-cavernosal injection of 100 unit of botulinum-A toxin plus daily intake of 5mg oral tadalafil in 32 adult diabetic patients with erectile dysfunction to detect its effect on on the erectile function status by reporting changes in IIEF and penile doppler parameters.

SECONDARY OUTCOMES:
Secondary adverse events of the drug. | 3months
  The second outcome is to assess the safety of the drug injection by reporting any secondary adverse events during or after injection such as mild pain, discomfort, edema, hematoma formation or chance of infection or psychological effects.

CONTACTS AND LOCATIONS:
Locations (1):
- Aswan University-Faculty of Medicine, Aswān, Aswan Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
Time Frame: starting 6-12 months after publication